CLINICAL TRIAL: NCT00727974
Title: Genetic Analysis of Children With Cyclic Vomiting Syndrome and Migraines
Brief Title: Genetic Analysis of Children With Cyclic Vomiting Syndrome (CVS) and Migraines
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Katja Kovacic, Professor of Gastroenterology, M.D., Medical College of Wisconsin
Other Study IDs: 08/24; GC 607
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Vomiting; Migraines
Keywords: Genome Wide Scan (GWS); Mitochondrial scan; Family trios
MeSH Terms: conditions — Vomiting; Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 ml of blood will be drawn through venipucture from the study subjects, their biological parents and siblings when available. In addition, 4 ml of blood will be drawn for serologic testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Diagnostic Criteria for CVS:
  3 or more different episodes of vomiting, normal health between episodes, no abnormal test results to account for vomiting [such as endoscopic biopsies (looking at a body part with a lighted tube), hydronephrosis (water block kidney drainage), cholelithiasis (gallstones), pancreatitis (swelling of the pancreas), and hypoglycemia (too little sugar in the blood)];
- 2: Diagnostic Criteria for Migraine:
  5 or more different headaches, complete return to health in between headaches, headaches last 2-48 hours and get in the way everyday activity, headache affects one side of head, with pounding moderate-to-severe pain, one of the following: nausea, vomiting, photophobia (fear of light), phonophobia (fear of sound).

SUMMARY:
The purpose of this study is to determine if there are genetic variations that can explain a genetic basis for cyclic vomiting syndrome (CVS).

DETAILED DESCRIPTION:
The purpose of this study is to determine if there are genetic variations that can explain a genetic basis for cyclic vomiting syndrome (CVS), various phenotypes of CVS (e.g. menstrual, Sato, calendar-tied) and migraine headaches (e.g. with aura, without aura, hemiplegic migraine). This information will allow physicians to improve care for patients who have been diagnosed with this disease and to provide their parents with more complete information regarding the cause of this disease. This research is being done because many unanswered questions remain regarding children with CVS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 0-21 years old with CVS (different phenotypes). Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent.

Exclusion Criteria:

* Subjects age > 22 years old Vomiting is not due to CVS or other related condition

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cyclic vomiting syndrome (CVS) may be the most severe recurrent vomiting disorder in humans. CVS is characterized by a sudden onset of rapid-fire vomiting, usually beginning in the early morning hours or upon wakening. It has a peak vomiting intensity of every 5-10 minutes (6-12 emeses) and episodes last between 2 hours and 10 days. These episodes of acute vomiting occur on average once every 2 to 4 weeks. The child returns to completely normal health between vomiting episodes. Children are diagnosed based on their specific vomiting pattern and a lack of positive findings on laboratory testing.
Sampling Method: Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2008-03-05 (Actual); Primary Completion 2013-06-12 (Actual); Study Completion 2013-06-12 (Actual)

PRIMARY OUTCOMES:
Identify novel genes that contribute to the risk of CVS using genomewide association analysis approach. | 3 years

SECONDARY OUTCOMES:
Perform genotype-phenotype correlations between genetic profiles and various phenotypes of CVS (e.g. menstrual, Sato, calendar-tied) and migraine headaches (e.g. with aura, without aura, hemiplegic migraine) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Katja Kovacic, MD, Principal Investigator — Medical College of Wiconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States